CLINICAL TRIAL: NCT05951842
Title: The Differences Between the Effects of Total Intravenous Anesthesia (TIVA) and Balanced Anesthesia on NK Cell and Cytokine Response in Colorectal Cancer Patients Undergoing Cytoreductive Surgery and HIPEC(Hyperthermic Intraperitoneal Chemotherapy)
Brief Title: Anesthesia, TIVA, Balanced Anesthesia, NK Cell
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: participants are no longer being examined or receiving intervention
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3-2017-0378
Record Dates: First submitted 2018-04-01; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA group (Active Comparator): In TIVA group, anesthesia will be maintained by propofol and remifentanil infusion under target controlled infusion.
  Other names: fresofol MCT 1% inj®; Fresenius kabi, Seoul, Korea, Ultian inj®; Hanlim, Seoul, Korea
  Interventions: Drug: anesthetic method
- Balanced anesthesia group. (Experimental): Anesthesia will be maintained by sevoflurane and remifentanil infusion in the balanced anesthesia group.
  Other names: Sojourn®, Kyongbo, Seoul, Korea, Ultian inj®; Hanlim, Seoul, Korea,
  Interventions: Drug: anesthetic method

INTERVENTIONS:
Drug: anesthetic method — Patients will be assigned to one of the groups, TIVA group or Balanced anesthesia group. In TIVA group, anesthesia will be maintained by propofol and remifentanil infusion under target controlled infusion. In contrast, anesthesia will be maintained by sevoflurane and remifentanil infusion in the balanced anesthesia group.

SUMMARY:
Anesthetic method was reported to have an impact on postoperative long-term outcome in cancer patients. In this study, we will investigate the effect of different anesthetic methods on NK cell activity, cytokine response and postoperative outcome in colorectal cancer patients undergoing CRS and HIPEC. We will compare propofol-based total intravenous anesthesia (TIVA) with balanced anesthesia to determine the effect of propofol, inhalation agent, and opioid on tumor genesis, recurrence, NK cell activity, cytokine response, and postoperative outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer patients undergoing elective cytoreductive surgery and HIPEC (20-70 yrs old)
2. American Society of Anesthesiologists physical status I, II, III

Exclusion Criteria:

1. Patients under 20 years old.
2. Patients with long-term steroid therapy or immunosuppressive therapy.
3. Patients with long-term NSAIDs therapy.
4. Patients who cannot communicate with other person or with cognitive disorder.
5. Patients who cannot read the consent form.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Postoperative immune function (NK cell count) | Postoperative day 1
  Postoperative immune function will be measured at baseline, POD#1, and POD#7. Postoperative immune function will be investigated by measuring NK cell count.

IPD SHARING:
Plan to Share IPD: No